CLINICAL TRIAL: NCT01027078
Title: Mechanism of Endothelial Dysfunction in Obstructive Sleep Apnea
Brief Title: Mechanism of Endothelial Dysfunction in Obstructive Sleep Apnea (OSA)
Status: Terminated | Type: Observational
Why Stopped: Due to insufficient grant funding
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: 2009H0212
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — skin biopsies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- OSA: patients diagnosed with obstructive sleep apnea who do not have existing cardiovascular disease
- control: patients without obstructive sleep apnea who are matched in weight and age to the OSA patients

SUMMARY:
The investigators hypothesized that patients with Obstructive Sleep Apnea (OSA) who are free of any cardiovascular disease will have early microcirculatory changes that are unique to OSA, and therefore would resolve with treatment of OSA.

DETAILED DESCRIPTION:
Impaired vascular regulation of the microcirculation is a consequence of Obstructive Sleep Apnea (OSA). Nitric Oxide (NO) related endothelial dysfunction occurs in OSA as the earliest vascular abnormality prior to the manifestation of vascular disease and it results in impaired vasodilatory response to hypoxia. These abnormalities have already been described in OSA patients. The role of oxidative stress in endothelial dysfunction is present in vascular disorders. The presence of oxidative stress in OSA patients is also well established. The effect of increased superoxide on endothelial function has also been described in the literature. The mechanism of this effect is unknown and is the focus of this research.

We hypothesized that patients with Obstructive Sleep Apnea (OSA) who are free of any cardiovascular disease will have early microcirculatory changes that are unique to OSA, and therefore would resolve with treatment of OSA.

ELIGIBILITY:
Inclusion criteria:

1. Apnea-Hypopnea Index (AHI) > 15 events per hours.

Exclusion criteria:

1. Hypertension defined by existing treatment with antihypertensives or any measurement of systolic pressure above 130 mmHg, or diastolic pressure above 85 mmHg;
2. Dyslipidemia defined by fasting cholesterol above 200; or fasting LDL over 150 mg/dl;
3. Diabetes defined as existing diagnosis, hemoglobin A1C >7 or fasting glucose >110 on two separate measurements (standard fasting glucose or HbA1C criteria);
4. CAD defined by history of angina, coronary event or abnormal stress test;
5. Peripheral Vascular Disease (PVD) defined by history of stroke, claudication or abnormal Ankle brachial index;
6. Concurrent smoking;
7. Pregnancy;
8. Use of erectile dysfunction drugs, or any medications for chronic conditions; 9)Chronic liver or renal disease. Fasting blood test for glucose, cholesterol, on all participants who have not had these tests in the 6 month prior to enrollment, will be obtained at the time of screening. The remaining criteria will be evaluated by reviewing the medical records and history taking on the day of first visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants: will be 36 patients with newly diagnosed OSA and 36 age and BMI matched controls.
  Patients with OSA will be enrolled from the sleep disorders center at OSU among patients who underwent a recent (past 4 weeks) polysomnography that is positive for OSA, and never were treated with CPAP.
  Inclusion criteria will be AHI > 15 events per hours.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
eNOS Expression | Measured at basline and 3-months post-treatment (CPAP) initiation
  All measurements will be obtained upon diagnosis of OSA and 12 weeks after effective treatment with continuous positive airway pressure (CPAP). Controls will receive all measurements at baseline.

SECONDARY OUTCOMES:
Peroxynitrite Formation | Measured at basline and 3-months post-treatment (CPAP) initiation
  All measurements will be obtained upon diagnosis of OSA and 12 weeks after effective treatment with continuous positive airway pressure (CPAP). Controls will receive all measurements at baseline.

OTHER OUTCOMES:
Superoxide Production | Measured at basline and 3-months post-treatment (CPAP) initiation
  All measurements will be obtained upon diagnosis of OSA and 12 weeks after effective treatment with continuous positive airway pressure (CPAP). Controls will receive all measurements at baseline.
Plasma BH2 and BH4 Levels | Measured at basline and 3-months post-treatment (CPAP) initiation
  All measurements will be obtained upon diagnosis of OSA and 12 weeks after effective treatment with continuous positive airway pressure (CPAP). Controls will receive all measurements at baseline. The BH2/BH4 ratio will be measured using high pressure liquid chromatography (HPLC).
Plasma ADMA Levels | Measured at basline and 3-months post-treatment (CPAP) initiation
  All measurements will be obtained upon diagnosis of OSA and 12 weeks after effective treatment with continuous positive airway pressure (CPAP). Controls will receive all measurements at baseline. Plasma ADMA levels will be measured using high pressure liquid chromatography (HPLC).

CONTACTS AND LOCATIONS:
Overall Officials: Rami Khayat, MD, Principal Investigator — Ohio State University
Locations (1):
- The Davis Heart and Lung Research Institute, Columbus, Ohio, United States